CLINICAL TRIAL: NCT02075944
Title: Effects of Aerobic Exercise on Cognitive Function and Brain-derived Neurotrophic Factor in Young Adults Aged 15-21 Years
Brief Title: Effects of Aerobic Exercise on Cognitive Function and Brain-derived Neurotrophic Factor in Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Southern Denmark (Other)
Responsible Party: Principal Investigator, Anna Bugge, Post Doc, PhD, University of Southern Denmark
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Supportive Care
Other Study IDs: S-20130171
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Physical Conditioning, Human; Cognition
Keywords: Aerobic exercise; Cognitive function; Executive function; Brain-derived neurotrophic factor
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High intensity aerobic exercise (Experimental): 30 minutes of high intensity aerobic exercise 3 times a weeks for 9 weeks - incorporation interval training
  Interventions: Behavioral: High intensity aerobic exercise
- Low intensity aerobic exercise (Experimental): 30 minutes of low intensity aerobic exercise 3 times a weeks for 9 weeks
  Interventions: Behavioral: Low intensity aerobic exercise
- Control (No Intervention): No intervention. Participants are told not to make any changes in their everyday life

INTERVENTIONS:
Behavioral: High intensity aerobic exercise
  Arms: High intensity aerobic exercise
Behavioral: Low intensity aerobic exercise
  Arms: Low intensity aerobic exercise

SUMMARY:
The present study will investigate the effects of aerobic exercise on cognition and growth factors including brain-derived neurotrophic factor (BDNF) in young adults aged 15-21 years. The included subjects will be randomized to three different groups including one control group and two exercise groups. Subjects randomized to the exercise groups will complete 30 minutes of aerobic exercise 3 times a week for 9 weeks incorporating low (group I) or high (group II) intensity aerobic exercise. The exercise will be conducted as running or indoor cycling (supervised). At baseline and 9-weeks follow-up all subjects will complete two cognitive tests (measures of concentration and sustained attention), a maximal cycling test (direct measures of VO2max), an intelligence quotient test, anthropometric measures, fasting blood samples and blood samples immediately following the cycling test. The blood samples will be analyzed for growth factors including BDNF and metabolic factors.

ELIGIBILITY:
Inclusion Criteria:

* age 15-21

Exclusion Criteria:

* injury preventing one from being physically active

Ages: 15 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 130 (Actual)
Dates: Start 2014-02; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The Flanker Task | 9 weeks
The AX-Continuous Performance test | 9 weeks
Brain-derived neurotrophic factor | 9 weeks

SECONDARY OUTCOMES:
Intelligence quotient | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Anne K Thorsen, Cand. Scient, Principal Investigator — University of Southern Denmark
Locations (1):
- University of Southern Denmark, Odense, Denmark

REFERENCES:
- [Derived] Gejl AK, Bugge A, Ernst MT, Mortensen EL, Gejl KD, Andersen LB. Effects of 9 Weeks of High- or Moderate-Intensity Training on Cardiorespiratory Fitness, Inhibitory Control, and Plasma Brain-Derived Neurotrophic Factor in Danish Adolescents-A Randomized Controlled Trial. Scand J Med Sci Sports. 2024 Aug;34(8):e14703. doi: 10.1111/sms.14703. PMID 39054765